CLINICAL TRIAL: NCT01142791
Title: A Phase IV Clinical Study To Evaluate the Safety of MR-Guided Focused Ultrasound Treatment of Uterine Fibroids With Enhanced Sonication Techniques
Brief Title: Safety Study of ExAblate for the Treatment of Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF033
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-01

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids; MRgFUS; ExAblate; Focused Ultrasound; Symptomatic uterine fibroids
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ExAblate treatment (Other)
  Interventions: Device: ExAblate

INTERVENTIONS:
Device: ExAblate — Magnetic resonance image-guided focused ultrasound (MRgFUS) for fibroid ablation

SUMMARY:
The objective of this Phase IV study is to evaluate the safety of the ExAblate treatment of uterine fibroids using the enhanced sonication techniques, based on the current commercially-approved treatment guidelines. Treatment may include up to 100% of individual fibroid volume, within established serosal and sacral treatment margins.

The Enhanced sonication is one of the various sonication modes that may lead to increased thermal dose volume of each sonication without additional safety risks. This is an additional treatment tool available in the ExAblate system for the treatment of uterine fibroids.

The safety profile of the Enhanced Sonication was investigated under an FDA-regulated IDE study. FDA granted approval of Enhanced Sonication with the requirement to perform a post-approval study to collect additional safety data when treating up to 100% of individual fibroid volume.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18 or older
* Symptomatic uterine fibroids, defined as those resulting in scores of 21 or higher, based on patient responses to questions 1-8 of the Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL)
* Women who have given written informed consent
* Women who are able and willing to attend all study visits.
* Patient is pre or peri-menopausal (within 12 months of last menstrual period).
* Patient should be family complete.
* Able to communicate sensations during the ExAblate procedure.
* Uterine fibroids, which are device accessible (i.e., positioned in the uterus such that they can be accessed without being shielded by bowel or bone).
* Fibroids(s) clearly visible on non-contrast MRI.
* Fibroid enhances on MR contrast imaging.

Exclusion Criteria:

* Women who are pregnant, as confirmed by serum/urine test at time of screening, or urine pregnancy test on the day of treatment.
* Patients who are breast-feeding.
* Patients with active pelvic inflammatory disease (PID).
* Patients with active local or systemic infection.
* Patients experiencing chronic leg or lower back pain within the last 6 months.
* Contraindication for MRI Scan:

  * Severe claustrophobia that would prevent completion of procedure in the MR unit
  * Weight greater than 250 lbs (113Kg)
  * Implanted ferromagnetic materials and/or devices contraindicated for MR scan
  * Known intolerance to MRI contrast agent (e.g. Gadolinium or Magnevist)
  * Any other contraindication for MRI Scan
* Extensive abdominal scarring in the beam path (that cannot be avoided by redirection of the beam).
* Dermoid cyst of the ovary anywhere in the treatment path.
* Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia.
* Intrauterine device (IUD) anywhere in the treatment path.
* Undiagnosed vaginal bleeding.
* Pedunculated fibroids.
* Uterine size >24 weeks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-05; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCLA, Los Angeles, California
  - UCSD Department of Radiology, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University Image Guided Therapy, Boca Raton, Florida
  - Borgess Research Institute, Kalamazoo, Michigan
  - Duke University, Durham, North Carolina
  - The Methodist Hospital Research Institute, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- See also: Sponsor's Web Page — http://www.insightec.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol defined the primary analysis to include participants receiving more than 1 sonication, i.e., 115 in this case. The safety population was defined in the protocol as participants receiving any sonications which is 121. 6 subjects receiving only 1 sonication were in the safety population but not in the baseline or primary analysis.
Groups:
- ExAblate Treatment: ExAblate: Magnetic resonance image-guided focused ultrasound (MRgFUS) for fibroid ablation. Phase IV enhanced sonication technique.
- Additional Safety Population Particpants: Per protocol 6 participants receiving only 1 sonication were added to the 115 ExAblate treated subjects to compose the full safety analysis population of 121. These 6 were included in adverse event reporting only, not in baseline or efficacy analyses.
Period: Overall Study
Arm/Group | ExAblate Treatment | Additional Safety Population Particpants
Started | 115 | 6 (6 participants receiving only 1 sonication were included only in adverse events reporting.)
Safety | 115 | 6 (Safety data only was reported for 6 participants receiving only 1 sonication.)
Completed | 108 | 0
Not Completed | 7 | 6
Not completed — Alternative Treatment | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Received only 1 sonication | 0 | 6

BASELINE CHARACTERISTICS:
Population: Baseline data is reported for the 115 participants who underwent the ExAblate treatment. Per protocol, 6 participants receiving only 1 sonication are included in the adverse events reporting only, not in the baseline or efficacy analyses..
Arm/Group | ExAblate Treatment
Number analyzed (Participants) | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  European/Middle East (White) | 84
  Hispanic | 6
  Black | 14
  Asian | 8
  Other | 3
Region of Enrollment [Number; unit: participants]
  United States | 115

OUTCOME MEASURES:

1. Primary Outcome: Percent Occurrence of Chronic Leg Pain
Description: The hypothesis was that over 90% of subjects would not experience chronic leg pain. A lower 95% Confidence Limit > 0.90 was considered statistically successful.
Time Frame: From treatment to 1-month post-treatment
Population: Per protocol the number of participants analyzed was the number of participants receiving more than one sonication. Six subjects receiving one sonication were excluded from the primary analysis but included in the safety population for a safety sample size n = 121.
Measure: Number (95% Confidence Interval); unit: percentage of subjects without leg pain
Arm/Group | ExAblate Treatment
Number analyzed (Participants) | 115
percentage of subjects without leg pain | 97 [92 to 99]

ADVERSE EVENTS:
Time Frame: 1 Month
Description: Per protocol a predetermined sample size of 115 participants receiving more than one sonication were included in the primary analysis. An additional 6 subjects receiving a single sonication were excluded from the primary analysis but included in the adverse events analysis for a safety sample size of 121.
Arm/Group | ExAblate Treatment
All-Cause Mortality (participants affected / at risk) | 0/121
Serious Adverse Events (participants affected / at risk) | 0/121
Other Adverse Events (participants affected / at risk) | 105/121
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Treatment (N=121)
Increased blood pressure (Vascular disorders) | 1 (1)
Erythema abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
Infection IV site (Skin and subcutaneous tissue disorders) | 1 (1)
Skin burn (Skin and subcutaneous tissue disorders) | 5 (5)
Skin pain sonication relaed (Surgical and medical procedures) | 54 (67)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Bloating abdomen (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1)
GI upset (Gastrointestinal disorders) | 1 (1)
Heartburn (Gastrointestinal disorders) | 2 (2)
Nausea/vomiting (Gastrointestinal disorders) | 11 (12)
Mass - fat necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramping position related (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramping muscle leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain neck/shoulder position related (Musculoskeletal and connective tissue disorders) | 3 (4)
Pubic bone soreness position related (Musculoskeletal and connective tissue disorders) | 1 (1)
Cramping muscle inguinal (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain lower extremity position related (Musculoskeletal and connective tissue disorders) | 14 (15)
Discomfort neck/shoulder position related (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenderness abdomen position related (Musculoskeletal and connective tissue disorders) | 1 (1)
Parasthesia (Nervous system disorders) | 2 (2)
Cramping Sonication related (Surgical and medical procedures) | 12 (12)
Cramping abdomen (General disorders) | 2 (2)
Cramping back/buttock/leg (General disorders) | 1 (1)
Pain uterine sonication related (Surgical and medical procedures) | 2 (2)
Discomfort back/buttock/leg sonication related (Surgical and medical procedures) | 1 (1)
Pain abdomen sonication related (Surgical and medical procedures) | 63 (78)
Pain back/buttock/leg sonication related (Surgical and medical procedures) | 70 (104)
Tenderness abdomen (General disorders) | 3 (3)
Edema/swelling abdome (Reproductive system and breast disorders) | 3 (4)
Amennorhia (Reproductive system and breast disorders) | 1 (1)
Cramping menstrual (Reproductive system and breast disorders) | 6 (6)
Vaginal discharge/bleeding (Reproductive system and breast disorders) | 7 (7)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 4 (4)
Flu (General disorders) | 1 (1)
Medication error (General disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Infection bladder (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 3 (3)
Cystitis (Renal and urinary disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No